CLINICAL TRIAL: NCT07403929
Title: Determination of the Effect of Fermented Grape Juice Consumption on Oxidative Stress and Inflammation Biomarkers and SIRT-1 Levels in Fibromyalgia Patients
Brief Title: The Effect of Fermented Grape Juice Consumption on Fibromyalgia Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuba Kahraman, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1422809
Record Dates: First submitted 2025-12-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia; Fibromyalgia (FM); Fibromyalgia Syndrome, Primary
Keywords: fibromyalgia; chronic pain; pain; inflammation; oxidative stress; sirtuin-1; SIRT1; gut microbiota; phytochemicals; nutrition
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Pain; Inflammation | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical Nutrition Therapy + Hardaliye (Experimental): Assigned Interventions:
  Medical Nutrition Therapy (MNT) Hardaliye (200 mL/day)
  Arm Description: Participants receive individualized MNT and consume 200 mL hardaliye once daily during the intervention period.
  Interventions: Behavioral: Medical Nutrition Therapy (MNT); Other: Hardaliye (200 mL/day)
- Medical Nutrition Therapy (Experimental): Assigned Interventions:
  Medical Nutrition Therapy (MNT) Arm Description: Participants receive individualized MNT; no study beverage is provided.
  Interventions: Behavioral: Medical Nutrition Therapy (MNT)
- Hardaliye (Experimental): Assigned Interventions:
  Hardaliye (200 mL/day) Arm Description: Participants consume 200 mL hardaliye once daily and continue usual diet; no MNT is provided.
  Interventions: Other: Hardaliye (200 mL/day)

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy (MNT) — Individually tailored medical nutrition therapy delivered using a standardized counseling framework, energy prescription derived from predictive equations and physical activity level, with standardized macronutrient targets and follow-up reinforcement per protocol.
  Arms: Medical Nutrition Therapy; Medical Nutrition Therapy + Hardaliye
Other: Hardaliye (200 mL/day) — Traditional grape-based fermented beverage dispensed in 200 mL bottles; participants consume 200 mL once daily for the intervention period with standardized intake instructions and product handling.
  Arms: Hardaliye; Medical Nutrition Therapy + Hardaliye

SUMMARY:
The goal of this clinical trial is to learn if a traditional grape-based fermented drink called hardaliye helps treat fibromyalgia in adult women. We will also learn whether adding hardaliye to a personalized nutrition plan works better than using either one alone.

The main questions are:

Does diet + hardaliye improve antioxidant status and lower oxidative stress more than diet only or hardaliye only? Does diet + hardaliye lower inflammation (TNF-α, IL-6, hs-CRP) and raise SIRT1 levels? Do these changes relate to less pain and better symptoms (fibromyalgia impact, gut symptoms, sleep, mood)? Are there benefits for weight, waist size, blood pressure, and blood lipids?

How the groups are compared:

Researchers will compare three groups for 8 weeks:

Diet + Hardaliye (personalized medical nutrition plan + one 200 mL bottle of hardaliye daily) Diet only (personalized medical nutrition plan) Hardaliye only (usual diet + one 200 mL bottle of hardaliye daily)

Participants will:

Drink one 200 mL bottle of hardaliye each day if assigned to Diet + Hardaliye or Hardaliye only Follow a personalized nutrition plan if assigned to Diet + Hardaliye or Diet only Visit the clinic at the start and end of the study, with brief check-ins around weeks 2, 4, and 6 Give blood samples before and after the 8-week period Complete short questionnaires on pain, fibromyalgia impact, gut symptoms, sleep, and mood Keep simple logs of daily drink intake and diet plan adherence, and report any side effects

Who can join:

Adult women (20-40 years) with doctor-diagnosed fibromyalgia and BMI 25.0-29.9 kg/m² who meet the study's health and medication criteria.

DETAILED DESCRIPTION:
This is a single-center, parallel-group, randomized clinical trial with three intervention conditions implemented over an 8-week period. After screening and baseline procedures, participants are assigned in a 1:1:1 ratio using a computer-generated block randomization sequence prepared by an independent researcher not otherwise involved in study conduct. Allocation concealment is maintained using sequentially numbered, opaque, sealed envelopes opened only after confirming eligibility.

Due to the dietary nature of the interventions, participant-level blinding is not feasible. However, biospecimen handling and laboratory analyses are performed on coded (anonymized) samples; laboratory personnel remain blinded to group assignment and time point to minimize measurement bias.

Personalized medical nutrition therapy (MNT) is delivered using a standardized counseling framework with individualized targets. Resting metabolic rate is estimated using the Mifflin-St Jeor equation, and daily energy prescription is derived using physical activity level (PAL). Macro-distribution targets are standardized (10-20% protein, 45-60% carbohydrate, 25-30% fat), with saturated fat <7% of energy and trans fat <1% to align with guidance-based cardiometabolic risk control.

To reduce confounding from background polyphenol exposure, participants are instructed to avoid high-polyphenol red/purple fruits and vegetables according to protocol-defined lists; diet plans are structured as three main meals plus 2-3 snacks, and standardized exchange lists are provided to support adherence.

Hardaliye intervention (product handling and quality assurance): The study beverage is sourced from a traditional producer in Kırklareli and manufactured via controlled spontaneous fermentation without starter culture.

Hardaliye is dispensed in 200 mL bottles and distributed weekly under cold-chain conditions; participants are instructed to consume the beverage daily within a consistent intake window (16:00-16:30) to standardize exposure timing.

To ensure batch-to-batch consistency, each production batch undergoes predefined acceptance checks (°Brix, pH, and titratable acidity), and key compositional markers are measured post-bottling (total phenolics via Folin-Ciocalteu, total monomeric anthocyanins via pH-differential method, and antioxidant capacity via ABTS-based TEAC). Analytical repeatability is monitored (replicates/parallel runs; CV target <10% with repeat testing if unmet).

Batches outside acceptance ranges (e.g., °Brix 20.5-21.8; pH 3.50-4.00; acidity 0.68-0.75 g/100 mL; and protocol-defined total phenolic/anthocyanin targets) are excluded from participant distribution.

Where relevant, chromatographic confirmation (HPLC-DAD) is used to verify the phenolic profile of the study product and support linkage of total phenolic estimates to compound-level composition.

Participants complete an initial screening visit followed by a baseline (Day 0) visit and an end-of-intervention (Week 8) visit, with brief interim check-ins at Weeks 2, 4, and 6 for adherence review and systematic safety monitoring. Interim contacts include beverage count/log review, reinforcement of dietary counseling where applicable, and adverse event solicitation/documentation.

Adherence is operationalized as ≥80% compliance with the assigned beverage intake and/or nutrition therapy targets; intake and adherence are captured using simple participant logs reviewed at each contact.

Dietary intake is assessed using structured food records collected at multiple time points (7-day records at baseline, Week 4, and Week 8; and additional 3-day records during specified weeks) to quantify energy and nutrient intake and to support adherence monitoring. Nutrient analyses are performed using BeBIS software and interpreted against national reference intakes.

Dietary polyphenol exposure is estimated using Phenol-Explorer (v3.6) to derive total polyphenols and relevant subclasses; an antioxidant diet quality score (DAQS) is calculated based on intake of key antioxidant nutrients. Physical activity is monitored via 24-hour recall on diary days, and PAL is derived using activity-specific PAR values combined with Mifflin-St Jeor BMR estimates to support stability of lifestyle exposure during follow-up.

Fasting venous blood is collected at baseline and Week 8 and processed according to institutional standard operating procedures (timing, centrifugation, aliquoting, storage). Samples are labeled with coded identifiers to preserve analytical blinding, and assays are performed following validated methods and kit instructions with internal QC steps documented prospectively.

Data are captured in structured case report forms and reconciled against visit checklists, distribution records, and participant logs. Primary analyses follow an intention-to-treat approach. Group differences in change over time are evaluated using repeated-measures modeling (e.g., linear mixed-effects models including group, time, and group×time interaction), with prespecified sensitivity analyses based on adherence and protocol deviations; missing-data handling and multiplicity procedures are defined in the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Female, 20-40 years
* BMI 25.0-29.9 kg/m²
* FM per 2016 ACR criteria; abdominal pain/cramp per SSS sub-item
* MEDAS ≤5 at screening.
* Willing to maintain habitual activity and comply with assigned intervention; able to provide informed consent.

Exclusion Criteria:

* Age <20 or >40
* BMI ≤24.99 or ≥30.0 kg/m²
* Professional athletes; night-shift workers
* Food allergies; acute infection; antibiotic use within past month or during intervention.
* Use (past 3 months) of dietary supplements; recent weight-loss or special diets (e.g., ketogenic).
* Pregnancy/lactation; menopause.
* Major hepatic/renal/cardiac/immune disease; chronic GI diseases; diabetes; CNS disorders; cancer; thyroid disease; severe pulmonary disease. Inflammatory arthritis/autoimmune disease impacting weight; medications including corticosteroids, estrogens, analgesics/anti-inflammatories, anti-diabetic or lipid-lowering drugs.
* Severe psychiatric illness/substance use; heavy alcohol/smoking.
* High recent intake of grape juice/molasses; excess tea/coffee (≥7 cups/day).
* Adherence <80% to beverage or MNT during run-in/screening.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients
Enrollment: 45 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised | Baseline to Week 8
  Change in FIQR (0-100); lower scores indicate less symptom burden and better function.
Pain Severity (Visual Analog Scale, VAS) | Baseline to Week 8
  Change in 0-10 cm VAS for average pain; lower scores reflect less pain.
Gastrointestinal symptoms (Gastrointestinal Symptom Rating Scale, GSRS) | Baseline to Week 8
  Change in Gastrointestinal Symptom Rating Scale (GSRS) total score and subscale scores (abdominal pain, reflux, diarrhea, dyspepsia/indigestion, constipation).
  The GSRS includes 15 items, each rated for the past week on a 7-point scale (1 = no discomfort, 7 = very severe discomfort). Higher scores indicate worse gastrointestinal symptoms and lower scores indicate fewer/milder symptoms.
  Total score (sum of 15 items): 15-105 Abdominal pain subscale (Items 1, 4, 5; sum): 3-21 Reflux subscale (Items 2, 3; sum): 2-14 Dyspepsia/Indigestion subscale (Items 6, 7, 8, 9; sum): 4-28 Diarrhea subscale (Items 11, 12, 14; sum): 3-21 Constipation subscale (Items 10, 13, 15; sum): 3-21
Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline to Week 8
  Change in PSQI global score (0-21); lower scores indicate better sleep quality.
Depressive Symptoms (Beck Depression Inventory, BDI) | Baseline to Week 8
  Change in BDI total score (0-63); lower scores indicate fewer depressive symptoms.

SECONDARY OUTCOMES:
Total Antioxidant Status (TAS; μmol Trolox eq/L) | Baseline to Week 8
  Change in circulating antioxidant capacity; higher values suggest stronger systemic antioxidant defense.
Total Oxidant Status (TOS; μmol H₂O₂ eq/L) | Baseline to Week 8
  Change in cumulative oxidant load; lower values indicate reduced oxidative pressure.
Oxidative Stress Index (OSI = TOS×100 / TAS) | Baseline to Week 8
  Ratio index of oxidant burden to antioxidant capacity; lower values denote better redox balance.
Plasma Malondialdehyde (MDA; TBARS method) | Baseline to Week 8
  Change in lipid peroxidation marker; lower levels indicate less oxidative membrane damage.
Serum 8-Hydroxy-2'-deoxyguanosine (8-OHdG) | Baseline to Week 8
  Change in DNA oxidative damage marker; lower concentrations suggest reduced nucleic acid oxidation.
Inflammatory biomarkers (TNF-α, IL-6, hs-CRP) | Baseline to Week 8
  Changes in systemic inflammation; reductions indicate attenuation of low-grade inflammatory activity.
Serum Sirtuin-1(SIRT1) | Baseline to Week 8
  Change in SIRT1 concentration (ELISA); higher levels are consistent with enhanced cellular stress-response signaling.

OTHER OUTCOMES:
Body Weight | Baseline to Week 8
  Body weight measured in light clothing without shoes using a calibrated scale. Units: kilograms (kg). Higher values indicate greater body mass.
Height | Baseline to Week 8
  Standing height measured without shoes using a calibrated stadiometer. Units: centimeters (cm). Height is collected primarily to compute BMI (kg/m²). Higher values indicate greater stature.
Body Mass Index (BMI) | Baseline to Week 8
  BMI calculated as weight (kg) / height (m²) using measured weight and height. Units: kg/m². Higher values indicate higher adiposity-related risk.
Waist Circumference | Baseline to Week 8
  Waist circumference measured at a standardized anatomical site using a non-elastic tape. Units: centimeters (cm). Higher values indicate greater central adiposity.
Waist-to-Hip Ratio (WHR) | Baseline to Week 8
  WHR calculated as waist circumference (cm) / hip circumference (cm) from standardized tape measurements. Units: ratio (unitless). Higher values indicate greater central fat distribution.
Systolic Blood Pressure (SBP) | Baseline to Week 8
  Seated systolic blood pressure measured after rest using a validated device per standardized procedure. Units: mmHg. Higher values indicate higher systolic pressure.
Diastolic Blood Pressure (DBP) | Baseline to Week 8
  Seated diastolic blood pressure measured after rest using a validated device per standardized procedure. Units: mmHg. Higher values indicate higher diastolic pressure.
Lipid Profile (total cholesterol, HDL-C, LDL-C, triglycerides) | Baseline to Week 8
  Changes indicate potential effects on atherogenic risk.
Dietary Polyphenol Intake (Phenol-Explorer-based total and subclasses) | Baseline to Week 8
  Estimated change in total/flavonoids/phenolic acids/flavanols/lignans; higher intake supports exposure to bioactive compounds.
Dietary Antioxidant Quality Score (DAQS) | Baseline to Week 8
  Description: Change in Dietary Antioxidant Quality Score (DAQS), a unitless composite score ranging from 0 to 5 derived from dietary intakes of vitamins A, C, and E, and the minerals zinc and selenium. For each nutrient, participants receive 1 point if their intake is ≥ 2/3 of the age- and sex-specific Recommended Dietary Allowance (RDA) / Dietary Reference Intake (DRI), and 0 points otherwise. Points are summed across the 5 nutrients (minimum 0, maximum 5). Higher DAQS indicates better dietary antioxidant quality (more adequate antioxidant-related nutrient intake), whereas lower scores indicate poorer dietary antioxidant quality.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Ayaz, Prof.Dr., Study Director — Hacettepe University Nutrition and Dietetics Department
Locations (1):
- İstanbul University-Cerrahpaşa Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I haven't started working on it yet and made progress.

REFERENCES:
- [Background] Erel O. A new automated colorimetric method for measuring total oxidant status. Clin Biochem. 2005 Dec;38(12):1103-11. doi: 10.1016/j.clinbiochem.2005.08.008. Epub 2005 Oct 7. PMID 16214125
- [Background] Erel O. A novel automated method to measure total antioxidant response against potent free radical reactions. Clin Biochem. 2004 Feb;37(2):112-9. doi: 10.1016/j.clinbiochem.2003.10.014. PMID 14725941
- [Background] Al-Aubaidy HA, Jelinek HF. Oxidative stress and triglycerides as predictors of subclinical atherosclerosis in prediabetes. Redox Rep. 2014 Mar;19(2):87-91. doi: 10.1179/1351000213Y.0000000080. Epub 2014 Jan 13. PMID 24520969
- [Background] Jentzsch AM, Bachmann H, Furst P, Biesalski HK. Improved analysis of malondialdehyde in human body fluids. Free Radic Biol Med. 1996;20(2):251-6. doi: 10.1016/0891-5849(95)02043-8. PMID 8746446
- [Background] Gerrior S, Juan W, Basiotis P. An easy approach to calculating estimated energy requirements. Prev Chronic Dis. 2006 Oct;3(4):A129. Epub 2006 Sep 15. PMID 16978504
- [Background] Bekar C, Goktas Z. Validation of the 14-item mediterranean diet adherence screener. Clin Nutr ESPEN. 2023 Feb;53:238-243. doi: 10.1016/j.clnesp.2022.12.026. Epub 2022 Dec 29. PMID 36657918
- [Background] Martinez-Gonzalez MA, Garcia-Arellano A, Toledo E, Salas-Salvado J, Buil-Cosiales P, Corella D, Covas MI, Schroder H, Aros F, Gomez-Gracia E, Fiol M, Ruiz-Gutierrez V, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Munoz MA, Warnberg J, Ros E, Estruch R; PREDIMED Study Investigators. A 14-item Mediterranean diet assessment tool and obesity indexes among high-risk subjects: the PREDIMED trial. PLoS One. 2012;7(8):e43134. doi: 10.1371/journal.pone.0043134. Epub 2012 Aug 14. PMID 22905215
- [Background] Rivas A, Romero A, Mariscal-Arcas M, Monteagudo C, Lopez G, Lorenzo ML, Ocana-Peinado FM, Olea-Serrano F. Association between dietary antioxidant quality score (DAQs) and bone mineral density in Spanish women. Nutr Hosp. 2012 Nov-Dec;27(6):1886-93. doi: 10.3305/nh.2012.27.6.6039. PMID 23588435
- [Background] Tur JA, Serra-Majem L, Romaguera D, Pons A. Does the diet of the Balearic population, a Mediterranean type diet, still provide adequate antioxidant nutrient intakes? Eur J Nutr. 2005 Jun;44(4):204-13. doi: 10.1007/s00394-004-0512-0. Epub 2004 Jul 7. PMID 15309419
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Ediz L, Hiz O, Toprak M, Tekeoglu I, Ercan S. The validity and reliability of the Turkish version of the Revised Fibromyalgia Impact Questionnaire. Clin Rheumatol. 2011 Mar;30(3):339-46. doi: 10.1007/s10067-010-1546-8. Epub 2010 Aug 12. PMID 20703890
- [Background] Sohrab G, Ebrahimof S, Sotoudeh G, Neyestani TR, Angoorani P, Hedayati M, Siasi F. Effects of pomegranate juice consumption on oxidative stress in patients with type 2 diabetes: a single-blind, randomized clinical trial. Int J Food Sci Nutr. 2017 Mar;68(2):249-255. doi: 10.1080/09637486.2016.1229760. Epub 2016 Sep 16. PMID 27633135
- [Background] Park M, Choi J, Lee HJ. Flavonoid-Rich Orange Juice Intake and Altered Gut Microbiome in Young Adults with Depressive Symptom: A Randomized Controlled Study. Nutrients. 2020 Jun 18;12(6):1815. doi: 10.3390/nu12061815. PMID 32570775
- [Background] Park YK, Lee SH, Park E, Kim JS, Kang MH. Changes in antioxidant status, blood pressure, and lymphocyte DNA damage from grape juice supplementation. Ann N Y Acad Sci. 2009 Aug;1171:385-90. doi: 10.1111/j.1749-6632.2009.04907.x. PMID 19723080
- [Background] Ghoochani N, Karandish M, Mowla K, Haghighizadeh MH, Jalali MT. The effect of pomegranate juice on clinical signs, matrix metalloproteinases and antioxidant status in patients with knee osteoarthritis. J Sci Food Agric. 2016 Oct;96(13):4377-81. doi: 10.1002/jsfa.7647. Epub 2016 Feb 22. PMID 26804926
- [Background] Martin KR , Burrell L , Bopp J . Authentic tart cherry juice reduces markers of inflammation in overweight and obese subjects: a randomized, crossover pilot study. Food Funct. 2018 Oct 17;9(10):5290-5300. doi: 10.1039/c8fo01492b. PMID 30255184
- [Background] Moynihan P, Makino Y, Petersen PE, Ogawa H. Implications of WHO Guideline on Sugars for dental health professionals. Community Dent Oral Epidemiol. 2018 Feb;46(1):1-7. doi: 10.1111/cdoe.12353. Epub 2017 Nov 23. PMID 29168887
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Casini I, Ladisa V, Clemente L, Delussi M, Rostanzo E, Peparini S, Aloisi AM, de Tommaso M. A Personalized Mediterranean Diet Improves Pain and Quality of Life in Patients with Fibromyalgia. Pain Ther. 2024 Jun;13(3):609-620. doi: 10.1007/s40122-024-00598-2. Epub 2024 Apr 29. PMID 38683449
- [Background] Castaldo G, Marino C, D'Elia M, Grimaldi M, Napolitano E, D'Ursi AM, Rastrelli L. The Effectiveness of the Low-Glycemic and Insulinemic (LOGI) Regimen in Maintaining the Benefits of the VLCKD in Fibromyalgia Patients. Nutrients. 2024 Nov 30;16(23):4161. doi: 10.3390/nu16234161. PMID 39683556
- [Background] Macian N, Duale C, Voute M, Leray V, Courrent M, Bode P, Giron F, Sonneville S, Bernard L, Joanny F, Menard K, Ducheix G, Pereira B, Pickering G. Short-Term Magnesium Therapy Alleviates Moderate Stress in Patients with Fibromyalgia: A Randomized Double-Blind Clinical Trial. Nutrients. 2022 May 17;14(10):2088. doi: 10.3390/nu14102088. PMID 35631229
- [Background] Baldi S, Pagliai G, Dinu M, Di Gloria L, Nannini G, Curini L, Pallecchi M, Russo E, Niccolai E, Danza G, Benedettelli S, Ballerini G, Colombini B, Bartolucci G, Ramazzotti M, Sofi F, Amedei A. Effect of ancient Khorasan wheat on gut microbiota, inflammation, and short-chain fatty acid production in patients with fibromyalgia. World J Gastroenterol. 2022 May 14;28(18):1965-1980. doi: 10.3748/wjg.v28.i18.1965. PMID 35664958
- [Background] Amoutzopoulos B, Loker GB, Samur G, Cevikkalp SA, Yaman M, Kose T, Pelvan E. Effects of a traditional fermented grape-based drink 'hardaliye' on antioxidant status of healthy adults: a randomized controlled clinical trial. J Sci Food Agric. 2013 Nov;93(14):3604-10. doi: 10.1002/jsfa.6158. Epub 2013 May 8. PMID 23553618
- [Background] Mittal M, Mehta P, Rajput S, Rajender S, Chattopadhyay N. The pharmacological assessment of resveratrol on preclinical models of rheumatoid arthritis through a systematic review and meta-analysis. Eur J Pharmacol. 2021 Nov 5;910:174504. doi: 10.1016/j.ejphar.2021.174504. Epub 2021 Sep 11. PMID 34520733
- [Background] Dani C, Dias KM, Trevizol L, Bassoa L, Fraga I, Proenca ICT, Pochmann D, Elsner VR. The impact of red grape juice (Vitis labrusca)consumption associated with physical training on oxidative stress, inflammatory and epigenetic modulation in healthy elderly women. Physiol Behav. 2021 Feb 1;229:113215. doi: 10.1016/j.physbeh.2020.113215. Epub 2020 Oct 21. PMID 33096120
- [Background] Choleva M, Argyrou C, Detopoulou M, Donta ME, Gerogianni A, Moustou E, Papaemmanouil A, Skitsa C, Kolovou G, Kalogeropoulos P, Fragopoulou E. Effect of Moderate Wine Consumption on Oxidative Stress Markers in Coronary Heart Disease Patients. Nutrients. 2022 Mar 25;14(7):1377. doi: 10.3390/nu14071377. PMID 35405991
- [Background] Fragopoulou E, Argyrou C, Detopoulou M, Tsitsou S, Seremeti S, Yannakoulia M, Antonopoulou S, Kolovou G, Kalogeropoulos P. The effect of moderate wine consumption on cytokine secretion by peripheral blood mononuclear cells: A randomized clinical study in coronary heart disease patients. Cytokine. 2021 Oct;146:155629. doi: 10.1016/j.cyto.2021.155629. Epub 2021 Jul 8. PMID 34247040
- [Background] Chiva-Blanch G, Urpi-Sarda M, Ros E, Valderas-Martinez P, Casas R, Arranz S, Guillen M, Lamuela-Raventos RM, Llorach R, Andres-Lacueva C, Estruch R. Effects of red wine polyphenols and alcohol on glucose metabolism and the lipid profile: a randomized clinical trial. Clin Nutr. 2013 Apr;32(2):200-6. doi: 10.1016/j.clnu.2012.08.022. Epub 2012 Sep 3. PMID 22999066
- [Background] Banini AE, Boyd LC, Allen JC, Allen HG, Sauls DL. Muscadine grape products intake, diet and blood constituents of non-diabetic and type 2 diabetic subjects. Nutrition. 2006 Nov-Dec;22(11-12):1137-45. doi: 10.1016/j.nut.2006.08.012. Epub 2006 Oct 9. PMID 17030113
- [Background] Aboutaleb AS, Allam A, Zaky HS, Harras MF, Farag FSA, Abdel-Sattar SA, El-Said NT, Ahmed HI, Abd El-Mordy FM. Novel insights into the molecular mechanisms underlying anti-nociceptive effect of myricitrin against reserpine-induced fibromyalgia model in rats: Implication of SIRT1 and miRNAs. J Ethnopharmacol. 2024 Dec 5;335:118623. doi: 10.1016/j.jep.2024.118623. Epub 2024 Jul 24. PMID 39059685
- [Background] Liou CJ, Wei CH, Chen YL, Cheng CY, Wang CL, Huang WC. Fisetin Protects Against Hepatic Steatosis Through Regulation of the Sirt1/AMPK and Fatty Acid beta-Oxidation Signaling Pathway in High-Fat Diet-Induced Obese Mice. Cell Physiol Biochem. 2018;49(5):1870-1884. doi: 10.1159/000493650. Epub 2018 Sep 20. PMID 30235452
- [Background] Singh A, Yadawa AK, Rizvi SI. Curcumin protects against aging-related stress and dysfunction through autophagy activation in rat brain. Mol Biol Rep. 2024 May 25;51(1):694. doi: 10.1007/s11033-024-09639-7. PMID 38796662
- [Background] Maleki MH, Abdizadeh Javazm S, Dastghaib S, Panji A, Hojjati Far M, Mahmoodi H, Siri M, Shafiee SM. The effect of quercetin on adipogenesis, lipolysis, and apoptosis in 3T3-L1 adipocytes: The role of SIRT1 pathways. Obes Sci Pract. 2024 Apr 13;10(2):e752. doi: 10.1002/osp4.752. eCollection 2024 Apr. PMID 38618521
- [Background] Garcia-Martinez BI, Ruiz-Ramos M, Pedraza-Chaverri J, Santiago-Osorio E, Mendoza-Nunez VM. Effect of Resveratrol on Markers of Oxidative Stress and Sirtuin 1 in Elderly Adults with Type 2 Diabetes. Int J Mol Sci. 2023 Apr 18;24(8):7422. doi: 10.3390/ijms24087422. PMID 37108584
- [Background] Brunet A, Sweeney LB, Sturgill JF, Chua KF, Greer PL, Lin Y, Tran H, Ross SE, Mostoslavsky R, Cohen HY, Hu LS, Cheng HL, Jedrychowski MP, Gygi SP, Sinclair DA, Alt FW, Greenberg ME. Stress-dependent regulation of FOXO transcription factors by the SIRT1 deacetylase. Science. 2004 Mar 26;303(5666):2011-5. doi: 10.1126/science.1094637. Epub 2004 Feb 19. PMID 14976264
- [Background] Ren Z, He H, Zuo Z, Xu Z, Wei Z, Deng J. The role of different SIRT1-mediated signaling pathways in toxic injury. Cell Mol Biol Lett. 2019 May 30;24:36. doi: 10.1186/s11658-019-0158-9. eCollection 2019. PMID 31164908
- [Background] Zhang H, Zhao Z, Pang X, Yang J, Yu H, Zhang Y, Zhou H, Zhao J. MiR-34a/sirtuin-1/foxo3a is involved in genistein protecting against ox-LDL-induced oxidative damage in HUVECs. Toxicol Lett. 2017 Aug 5;277:115-122. doi: 10.1016/j.toxlet.2017.07.216. Epub 2017 Jul 5. PMID 28688900
- [Background] Singh CK, Chhabra G, Ndiaye MA, Garcia-Peterson LM, Mack NJ, Ahmad N. The Role of Sirtuins in Antioxidant and Redox Signaling. Antioxid Redox Signal. 2018 Mar 10;28(8):643-661. doi: 10.1089/ars.2017.7290. Epub 2017 Oct 20. PMID 28891317
- [Background] Iside C, Scafuro M, Nebbioso A, Altucci L. SIRT1 Activation by Natural Phytochemicals: An Overview. Front Pharmacol. 2020 Aug 7;11:1225. doi: 10.3389/fphar.2020.01225. eCollection 2020. PMID 32848804
- [Background] Wong A, Woodcock EA. FoxO proteins and cardiac pathology. Adv Exp Med Biol. 2009;665:78-89. doi: 10.1007/978-1-4419-1599-3_6. PMID 20429417
- [Background] Yeung AWK, Tzvetkov NT, El-Tawil OS, Bungau SG, Abdel-Daim MM, Atanasov AG. Antioxidants: Scientific Literature Landscape Analysis. Oxid Med Cell Longev. 2019 Jan 8;2019:8278454. doi: 10.1155/2019/8278454. eCollection 2019. PMID 30728893
- [Background] Rodgers JT, Lerin C, Haas W, Gygi SP, Spiegelman BM, Puigserver P. Nutrient control of glucose homeostasis through a complex of PGC-1alpha and SIRT1. Nature. 2005 Mar 3;434(7029):113-8. doi: 10.1038/nature03354. PMID 15744310
- [Background] Kauppinen A, Suuronen T, Ojala J, Kaarniranta K, Salminen A. Antagonistic crosstalk between NF-kappaB and SIRT1 in the regulation of inflammation and metabolic disorders. Cell Signal. 2013 Oct;25(10):1939-48. doi: 10.1016/j.cellsig.2013.06.007. Epub 2013 Jun 11. PMID 23770291
- [Background] Wicinski M, Erdmann J, Nowacka A, Kuzminski O, Michalak K, Janowski K, Ohla J, Biernaciak A, Szambelan M, Zabrzynski J. Natural Phytochemicals as SIRT Activators-Focus on Potential Biochemical Mechanisms. Nutrients. 2023 Aug 14;15(16):3578. doi: 10.3390/nu15163578. PMID 37630770
- [Background] Yu X, Zhang S, Zhao D, Zhang X, Xia C, Wang T, Zhang M, Liu T, Huang W, Wu B. SIRT1 inhibits apoptosis in in vivo and in vitro models of spinal cord injury via microRNA-494. Int J Mol Med. 2019 Apr;43(4):1758-1768. doi: 10.3892/ijmm.2019.4106. Epub 2019 Feb 22. PMID 30816451
- [Background] Zhou C, Wu Y, Ding X, Shi N, Cai Y, Pan ZZ. SIRT1 Decreases Emotional Pain Vulnerability with Associated CaMKIIalpha Deacetylation in Central Amygdala. J Neurosci. 2020 Mar 11;40(11):2332-2342. doi: 10.1523/JNEUROSCI.1259-19.2020. Epub 2020 Jan 31. PMID 32005763
- [Background] O'Callaghan C, Vassilopoulos A. Sirtuins at the crossroads of stemness, aging, and cancer. Aging Cell. 2017 Dec;16(6):1208-1218. doi: 10.1111/acel.12685. Epub 2017 Oct 10. PMID 28994177
- [Background] Waldman M, Cohen K, Yadin D, Nudelman V, Gorfil D, Laniado-Schwartzman M, Kornwoski R, Aravot D, Abraham NG, Arad M, Hochhauser E. Regulation of diabetic cardiomyopathy by caloric restriction is mediated by intracellular signaling pathways involving 'SIRT1 and PGC-1alpha'. Cardiovasc Diabetol. 2018 Aug 2;17(1):111. doi: 10.1186/s12933-018-0754-4. PMID 30071860
- [Background] Haigis MC, Sinclair DA. Mammalian sirtuins: biological insights and disease relevance. Annu Rev Pathol. 2010;5:253-95. doi: 10.1146/annurev.pathol.4.110807.092250. PMID 20078221
- [Background] Chang HC, Guarente L. SIRT1 and other sirtuins in metabolism. Trends Endocrinol Metab. 2014 Mar;25(3):138-45. doi: 10.1016/j.tem.2013.12.001. Epub 2013 Dec 30. PMID 24388149
- [Background] Pagliai G, Giangrandi I, Dinu M, Sofi F, Colombini B. Nutritional Interventions in the Management of Fibromyalgia Syndrome. Nutrients. 2020 Aug 20;12(9):2525. doi: 10.3390/nu12092525. PMID 32825400
- [Background] Badaeva A, Danilov A, Kosareva A, Lepshina M, Novikov V, Vorobyeva Y, Danilov A. Neuronutritional Approach to Fibromyalgia Management: A Narrative Review. Pain Ther. 2024 Oct;13(5):1047-1061. doi: 10.1007/s40122-024-00641-2. Epub 2024 Jul 23. PMID 39042252
- [Background] Tel Adiguzel K, Koroglu O, Yasar E, Tan AK, Samur G. The relationship between dietary total antioxidant capacity, clinical parameters, and oxidative stress in fibromyalgia syndrome: A novel point of view. Turk J Phys Med Rehabil. 2022 Jun 1;68(2):262-270. doi: 10.5606/tftrd.2022.9741. eCollection 2022 Jun. PMID 35989949
- [Background] Fernandez-Araque A, Verde Z, Torres-Ortega C, Sainz-Gil M, Velasco-Gonzalez V, Gonzalez-Bernal JJ, Mielgo-Ayuso J. Effects of Antioxidants on Pain Perception in Patients with Fibromyalgia-A Systematic Review. J Clin Med. 2022 Apr 27;11(9):2462. doi: 10.3390/jcm11092462. PMID 35566585
- [Background] Kadayifci FZ, Bradley MJ, Onat AM, Shi HN, Zheng S. Review of nutritional approaches to fibromyalgia. Nutr Rev. 2022 Nov 7;80(12):2260-2274. doi: 10.1093/nutrit/nuac036. PMID 35674686
- [Background] Maddox EK, Massoni SC, Hoffart CM, Takata Y. Dietary Effects on Pain Symptoms in Patients with Fibromyalgia Syndrome: Systematic Review and Future Directions. Nutrients. 2023 Jan 31;15(3):716. doi: 10.3390/nu15030716. PMID 36771421
- [Background] Hauser W, Thieme K, Turk DC. Guidelines on the management of fibromyalgia syndrome - a systematic review. Eur J Pain. 2010 Jan;14(1):5-10. doi: 10.1016/j.ejpain.2009.01.006. Epub 2009 Mar 4. PMID 19264521
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Walitt B, Nahin RL, Katz RS, Bergman MJ, Wolfe F. The Prevalence and Characteristics of Fibromyalgia in the 2012 National Health Interview Survey. PLoS One. 2015 Sep 17;10(9):e0138024. doi: 10.1371/journal.pone.0138024. eCollection 2015. PMID 26379048
- [Background] Cabo-Meseguer A, Cerda-Olmedo G, Trillo-Mata JL. Fibromyalgia: Prevalence, epidemiologic profiles and economic costs. Med Clin (Barc). 2017 Nov 22;149(10):441-448. doi: 10.1016/j.medcli.2017.06.008. Epub 2017 Jul 19. English, Spanish. PMID 28734619
- [Background] Queiroz LP. Worldwide epidemiology of fibromyalgia. Curr Pain Headache Rep. 2013 Aug;17(8):356. doi: 10.1007/s11916-013-0356-5. PMID 23801009
- [Background] Schulze NBB, Barreto TDNP, Alencar GG, da Silva TA, Duarte ALBP, Ranzolin A, Siqueira GR. The effect of myofascial release of the physiological chains on the pain and health status in patients with fibromyalgia, compared to passive muscle stretching and a control group: a randomized controlled clinical trial. Disabil Rehabil. 2024 Aug;46(16):3629-3642. doi: 10.1080/09638288.2023.2255130. Epub 2023 Sep 12. PMID 37698013
- [Background] Fonseca ACS, Faria PC, Alcantara MA, Pinto WD, De Carvalho LG, Lopes FG, Pernambuco AP. Effects of aquatic physiotherapy or health education program in women with fibromyalgia: a randomized clinical trial. Physiother Theory Pract. 2021 May;37(5):620-632. doi: 10.1080/09593985.2019.1639229. Epub 2019 Jul 15. PMID 31305209
- [Background] Beck AT, Guth D, Steer RA, Ball R. Screening for major depression disorders in medical inpatients with the Beck Depression Inventory for Primary Care. Behav Res Ther. 1997 Aug;35(8):785-91. doi: 10.1016/s0005-7967(97)00025-9. PMID 9256522
- [Background] Kleykamp BA, Ferguson MC, McNicol E, Bixho I, Arnold LM, Edwards RR, Fillingim R, Grol-Prokopczyk H, Turk DC, Dworkin RH. The Prevalence of Psychiatric and Chronic Pain Comorbidities in Fibromyalgia: an ACTTION systematic review. Semin Arthritis Rheum. 2021 Feb;51(1):166-174. doi: 10.1016/j.semarthrit.2020.10.006. Epub 2020 Dec 29. PMID 33383293
- [Background] Magni G, Marchetti M, Moreschi C, Merskey H, Luchini SR. Chronic musculoskeletal pain and depressive symptoms in the National Health and Nutrition Examination. I. Epidemiologic follow-up study. Pain. 1993 May;53(2):163-168. doi: 10.1016/0304-3959(93)90076-2. PMID 8336986
- [Background] Chang MH, Hsu JW, Huang KL, Su TP, Bai YM, Li CT, Yang AC, Chang WH, Chen TJ, Tsai SJ, Chen MH. Bidirectional Association Between Depression and Fibromyalgia Syndrome: A Nationwide Longitudinal Study. J Pain. 2015 Sep;16(9):895-902. doi: 10.1016/j.jpain.2015.06.004. Epub 2015 Jun 25. PMID 26117813
- [Background] Berwick R, Barker C, Goebel A; guideline development group. The diagnosis of fibromyalgia syndrome. Clin Med (Lond). 2022 Nov;22(6):570-574. doi: 10.7861/clinmed.2022-0402. PMID 36427885
- [Background] National Guideline Centre (UK). Evidence review for pain management programmes for chronic pain (chronic primary pain and chronic secondary pain): Chronic pain (primary and secondary) in over 16s: assessment of all chronic pain and management of chronic primary pain: Evidence review C. London: National Institute for Health and Care Excellence (NICE); 2021 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK569980/ PMID 33939361
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Osorio CD, Gallinaro AL, Lorenzi-Filho G, Lage LV. Sleep quality in patients with fibromyalgia using the Pittsburgh Sleep Quality Index. J Rheumatol. 2006 Sep;33(9):1863-5. Epub 2006 Aug 15. PMID 16924687
- [Background] Martinez-Rodriguez A, Rubio-Arias JA, Ramos-Campo DJ, Reche-Garcia C, Leyva-Vela B, Nadal-Nicolas Y. Psychological and Sleep Effects of Tryptophan and Magnesium-Enriched Mediterranean Diet in Women with Fibromyalgia. Int J Environ Res Public Health. 2020 Mar 26;17(7):2227. doi: 10.3390/ijerph17072227. PMID 32224987
- [Background] Aslan CIn NN, Acik M, TertemIz OF, Aktan C, Akcali DT, Cakiroglu FP, OzcelIk AO. Effect of prebiotic and probiotic supplementation on reduced pain in patients with fibromyalgia syndrome: a double-blind, placebo-controlled randomized clinical trial. Psychol Health Med. 2024 Mar;29(3):528-541. doi: 10.1080/13548506.2023.2216464. Epub 2023 May 24. PMID 37224267
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Choy EH. The role of sleep in pain and fibromyalgia. Nat Rev Rheumatol. 2015 Sep;11(9):513-20. doi: 10.1038/nrrheum.2015.56. Epub 2015 Apr 28. PMID 25907704
- [Background] Gupte PA, Mahajan MP, Revadkar Kole MS, Mandlecha AH, Tatke PA, Naharwar VA, Bhalerao SS. Efficacy and acceptability of pomegranate effervescent granules in patients suffering from acid peptic disorders. Indian J Pharmacol. 2022 Jan-Feb;54(1):7-12. doi: 10.4103/ijp.ijp_914_20. PMID 35343201
- [Background] Junghard O, Wiklund IK. Effect of baseline symptom severity on patient-reported outcomes in gastroesophageal reflux disease. Eur J Gastroenterol Hepatol. 2007 Jul;19(7):555-60. doi: 10.1097/MEG.0b013e328133f2d1. PMID 17556901
- [Background] Hata S, Nakajima H, Hashimoto Y, Miyoshi T, Hosomi Y, Okamura T, Majima S, Nakanishi N, Senmaru T, Osaka T, Okada H, Ushigome E, Hamaguchi M, Asano M, Yamazaki M, Fukui M. Effects of probiotic Bifidobacterium bifidum G9-1 on the gastrointestinal symptoms of patients with type 2 diabetes mellitus treated with metformin: An open-label, single-arm, exploratory research trial. J Diabetes Investig. 2022 Mar;13(3):489-500. doi: 10.1111/jdi.13698. Epub 2021 Nov 15. PMID 34665938
- [Background] Wright-McNaughton M, Ten Bokkel Huinink S, Frampton CMA, McCombie AM, Talley NJ, Skidmore PML, Gearry RB. Measuring Diet Intake and Gastrointestinal Symptoms in Irritable Bowel Syndrome: Validation of the Food and Symptom Times Diary. Clin Transl Gastroenterol. 2019 Dec;10(12):e00103. doi: 10.14309/ctg.0000000000000103. PMID 31800544
- [Background] Remes-Troche JM, Taboada-Liceaga H, Gill S, Amieva-Balmori M, Rossi M, Hernandez-Ramirez G, Garcia-Mazcorro JF, Whelan K. Nopal fiber (Opuntia ficus-indica) improves symptoms in irritable bowel syndrome in the short term: a randomized controlled trial. Neurogastroenterol Motil. 2021 Feb;33(2):e13986. doi: 10.1111/nmo.13986. Epub 2020 Sep 16. PMID 32935904
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Background] Erdrich S, Hawrelak JA, Myers SP, Harnett JE. A systematic review of the association between fibromyalgia and functional gastrointestinal disorders. Therap Adv Gastroenterol. 2020 Dec 8;13:1756284820977402. doi: 10.1177/1756284820977402. eCollection 2020. PMID 33343707
- [Background] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Background] Gifford RW Jr. The arteriospastic diseases: clinical significance and management. Cardiovasc Clin. 1971;3(1):127-39. No abstract available. PMID 5119830
- [Background] D'Onghia M, Ciaffi J, Lisi L, Mancarella L, Ricci S, Stefanelli N, Meliconi R, Ursini F. Fibromyalgia and obesity: A comprehensive systematic review and meta-analysis. Semin Arthritis Rheum. 2021 Apr;51(2):409-424. doi: 10.1016/j.semarthrit.2021.02.007. Epub 2021 Mar 3. PMID 33676126
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Shukla V, Kumar DS, Ali MA, Agarwal S, Khandpur S. Nitric oxide, lipid peroxidation products, and antioxidants in primary fibromyalgia and correlation with disease severity. J Med Biochem. 2020 Jan 23;39(2):165-170. doi: 10.2478/jomb-2019-0033. PMID 33033448
- [Background] Andrade A, Vilarino GT, Sieczkowska SM, Coimbra DR, Steffens RAK, Vietta GG. Acute effects of physical exercises on the inflammatory markers of patients with fibromyalgia syndrome: A systematic review. J Neuroimmunol. 2018 Mar 15;316:40-49. doi: 10.1016/j.jneuroim.2017.12.007. Epub 2017 Dec 12. PMID 29254627
- [Background] O'Mahony LF, Srivastava A, Mehta P, Ciurtin C. Is fibromyalgia associated with a unique cytokine profile? A systematic review and meta-analysis. Rheumatology (Oxford). 2021 Jun 18;60(6):2602-2614. doi: 10.1093/rheumatology/keab146. PMID 33576773
- [Background] Dos Santos JM, Rodrigues Lacerda AC, Ribeiro VGC, Scheidt Figueiredo PH, Fonseca SF, da Silva Lage VK, Costa HS, Pereira Lima V, Sanudo B, Bernardo-Filho M, da Cunha de Sa Caputo D, Mendonca VA, Taiar R. Oxidative Stress Biomarkers and Quality of Life Are Contributing Factors of Muscle Pain and Lean Body Mass in Patients with Fibromyalgia. Biology (Basel). 2022 Jun 19;11(6):935. doi: 10.3390/biology11060935. PMID 35741454
- [Background] Assavarittirong C, Samborski W, Grygiel-Gorniak B. Oxidative Stress in Fibromyalgia: From Pathology to Treatment. Oxid Med Cell Longev. 2022 Oct 5;2022:1582432. doi: 10.1155/2022/1582432. eCollection 2022. PMID 36246401
- [Background] Ovrom EA, Mostert KA, Khakhkhar S, McKee DP, Yang P, Her YF. A Comprehensive Review of the Genetic and Epigenetic Contributions to the Development of Fibromyalgia. Biomedicines. 2023 Apr 7;11(4):1119. doi: 10.3390/biomedicines11041119. PMID 37189737
- [Background] Di Franco M, Iannuccelli C, Valesini G. Neuroendocrine immunology of fibromyalgia. Ann N Y Acad Sci. 2010 Apr;1193:84-90. doi: 10.1111/j.1749-6632.2009.05344.x. PMID 20398012
- [Background] Mahdi AA, Fatima G. A quest for better understanding of biochemical changes in fibromyalgia syndrome. Indian J Clin Biochem. 2014 Jan;29(1):1-2. doi: 10.1007/s12291-013-0395-z. Epub 2013 Nov 20. No abstract available. PMID 24478541
- [Background] Ghafouri B, Matikhan D, Christidis N, Ernberg M, Kosek E, Mannerkorpi K, Gerdle B, Wahlen K. The Vastus Lateralis Muscle Interstitium Proteome Changes after an Acute Nociception in Patients with Fibromyalgia Compared to Healthy Subjects-A Microdialysis Study. Biomedicines. 2023 Jan 13;11(1):206. doi: 10.3390/biomedicines11010206. PMID 36672714
- [Background] Jurado-Priego LN, Cueto-Urena C, Ramirez-Exposito MJ, Martinez-Martos JM. Fibromyalgia: A Review of the Pathophysiological Mechanisms and Multidisciplinary Treatment Strategies. Biomedicines. 2024 Jul 11;12(7):1543. doi: 10.3390/biomedicines12071543. PMID 39062116

DOCUMENTS (2):
  • Study Protocol (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT07403929/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT07403929/SAP_001.pdf